CLINICAL TRIAL: NCT02924025
Title: Motivational Interviewing as an Intervention for Women With Polycystic Ovary Syndrome and BMI Above 30 kg/m2
Brief Title: Motivational Interviewing as an Intervention for PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Pernille Ravn, Doktor med., Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Motivational interviewing PCOS
Record Dates: First submitted 2014-09-25; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Polycystic Ovary Syndrome; Overweight and Obesity; Motivation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case (Experimental): The women in this group will receive motivational interviews approximately once every 2 weeks for half a year.
  Interventions: Behavioral: Motivational interview
- Control (No Intervention): The women in this group will have the usual guidance in weightloss with a booklet on the seven health tips from the danish government. They will not be contacted ind the half year between study onset and finish.

INTERVENTIONS:
Behavioral: Motivational interview — Motivational interview is an interview form based on the patients own thoughts of motivation. It will be conducted by a nurse who is specially trained in this interview type.
  Arms: Case

SUMMARY:
The aim of the study is to examine if motivational interviewing can have a positive effect on weight loss over a 6 month period. By losing weight, the investigators assume the patients will have a positive effect on quality of life, and also that weight loss will help to regulate the factors that are present with polycystic ovary syndrom (PCOS); such as menstrual disorders and infertility.

Participants will be randomly assigned to a treatment group and a control group.

Both groups will be followed as normal with blood samples and other tests such as scans of the ovaries and measurement of height and weight at the beginning of the study and after six months.

In addition, there will be a small hair sample taken from the neck at the first consultation and after 6 months. This is done to measure the stress hormone cortisol in the body over the duration of the experiment.

The treatment group receive individual motivational interviews by a nurse every 14 days for a period of six months. After half a year, tests are repeated to see if there are significant differences between the groups.

DETAILED DESCRIPTION:
Main Hypothesis: Overweight women with PCOS receiving motivational interviewing lose at least 1.5 kg more than the control group during the 6 months.

Hypothesis: weight loss leads to positive changes in biochemical parameters, quality of life, and the stress levels assessed by cortisol levels in hair.

Research Plan:

The project began on october 1, 2014 at Odense University Hospital, gynecological and obstetric department. Women referred to the gynecology outpatient clinic for examination of PCOS was examined in the gynecological clinic at the appointment. The women who subsequently are diagnosed with PCOS and have a BMI> 30 kg/m2, who said yes to participation in the trial was randomized to motivational interviews or normal course of treatment.

Both groups: questionnaires and hair samples in both randomized groups. The investigators take about 150 strands of hair of 3 cm length twice in the experiment. Attendance for Biochemistry and objective examinations like the usual procedures for patients with PCOS, ie. this is performed whether the patient is involved in the trial or not. There will be two blood counts during the experiment, one at the start and one at 6 months. Blood sampling is carried out whether the patient is involved in the trial or not. Parameters measured at baseline and after 6 months:

Study program as usual (all patients with PCOS):

* anamneses of menstruation, fertility, use of oral contraceptives, medicine and disease ect.
* anthropometry: height, weight, body mass index (BMI), waist and hip circumference. Blood pressure.
* Biochemistry: fasting blood glucose, HbA1c, insulin, Lutropin hormone (LH), folicle stimulation hormone (FSH), estradiol, free and total testosterone,dehydroepiandrosteron (DHEAS),sex hormon binding globulin (SHBG), prolactin, thyroid stimulating hormone (TSH), 17-OH-progesterone, lipid profile, hemoglobin, 25-OH vitamin D.
* gynecological assessment: Ultrasound scanning of the uterus and ovaries.

Project participants:

* Questionnaires; SF-36, VAS score, major depression score (MDI), the world health organization WHO-five well-being index.
* hair sample for the detection of cortisol

Practical course:

First examination in the clinic: If the patient meets the inclusion criteria an in-depth information about the trial is given. If the patient wants to participate, the patient is issued a written statement of consent and is pre booked an appointment with a nurse At the first visit to the nurse: the consent form is signed, if wish for participation in the study is maintained the patient is randomized. The patient fill out questionnaires and a hair sample is taken. All patients are provided with information on weight loss from the Health Protection Agency advice about diet and exercise as above. Patients who are randomized to motivational interviews starts a course of interviews. Participant data is imported into a spreadsheet for later determination.

Intervention: appointments of interview are scheduled individually, but should be around one interview every 14 days of about 20 minutes.

After 6 months, all patients are examined again as mentioned above as part of the usual control of PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Women with polycystic ovary syndrome and BMI above 30 kg/m2

Exclusion Criteria:

* Women taking gender hormone medication, for example birthcontrol pills.
* Metformin treatment in less than 3 months (i.e. women who is in a stable treatment and have been taking metformin in more than 3 months, is allowed to participate)
* women who can not read/understand danish, and is in need of a translater.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months
  Measured as change in kg, body mass index and hip to waist circumference

SECONDARY OUTCOMES:
Quality of life | 6 months
  Assessed by questionnaires: WHO five score, major depression index, a VAS score of 10 and a PCOS questionnaire.
Less symptoms of PCOS | 6 months
  Measured in change in androgen hair growth of body and face, menstruation, acne, pain, hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Ravn, MD, Study Chair — Department of Gynocology and obstetrics D, Odense University Hospital

IPD SHARING:
Plan to Share IPD: Yes
The plan is to publish the results by the end of 2016. Individual participant data will be available by request

REFERENCES:
- [Derived] Moeller LV, Lindhardt CL, Andersen MS, Glintborg D, Ravn P. Motivational interviewing in obese women with polycystic ovary syndrome - a pilot study. Gynecol Endocrinol. 2019 Jan;35(1):76-80. doi: 10.1080/09513590.2018.1498832. Epub 2018 Sep 5. PMID 30182773